CLINICAL TRIAL: NCT05241379
Title: Exploratory Safety and Electrophysiological Study of Closed-loop Pudendal Neuromodulation Using an Implantable (Picostim-DyNeuMo) Device in Women With Urinary Incontinence
Brief Title: AURA-2: Augmenting Urinary Reflex Activity
Acronym: AURA-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amber Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Amber AURA-2
Record Dates: First submitted 2022-01-24; First posted 2022-02-15 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Overactive Bladder; Urge Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amber UI Therapy (Experimental): Participants will undergo surgical implantation of the Amber UI System incorporating 2 electrode leads connected to a single IPG
  Interventions: Device: Amber UI System

INTERVENTIONS:
Device: Amber UI System — The implantable components of the Amber UI system consist of an implantable pulse generator (Picostim Amber IPG), 2 electrode leads with anchoring system

SUMMARY:
AMBER AURA-2 study (Augmenting Urinary Reflex Activity 2) is a short-duration (6 month) safety and electrophysiological study using an implanted Amber UI system and two electrode leads to provide closed-loop pudendal nerve stimulation for the treatment of urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥ 18 years
* Diagnosis of urinary incontinence, with on a 5-day voiding diary at least 1 daily urgency episode and/or greater than or equal to 8 voids/day and/or by having a minimum of two involuntary leaking episodes in 72 hr
* Duration of urinary incontinence symptom ≥ 6 months prior to the screening baseline visit date
* Failed or is not a candidate for more conservative treatment e.g. pelvic floor muscle therapy or biofeedback or behavioral modification
* Failed or could not tolerate at least one (1) antimuscarinic or beta3-adrenoceptor agonist medication
* Urodynamic testing (uroflowmetry, cystometry and pressure flow) completed within 12 months prior to screening baseline visit date or is willing to have testing at screening baseline visit
* Cystoscopy test completed within 12 months prior to the screening baseline visit date or is willing to have a test at screening baseline visit
* Is willing and able to washout from OAB medications for at least 4 week prior to beginning the baseline voiding diary
* Ability and willingness to give informed consent including language constraints (see above)
* Able to participate in all testing and follow-up clinic visits associated with study protocol
* Capable of independently using the system components (after training) as described in the Patient Manual
* Mobile and able to use toilet without assistance

Exclusion Criteria:

General:

* Patient is pregnant, breastfeeding, or plans to become pregnant during the course of the study (pregnancy tests provided in schedule)
* Patient is unwilling or unable to use contraception during sexual intercourse for the duration of the study, and thereafter if implant remains in the longer term.
* Any significant medical condition that is likely to interfere with study procedures, device operation, or likely to confound evaluation of study endpoints
* Any psychiatric or personality disorder at the discretion of the study physician
* Any neurological condition that may interfere with normal bladder function (e.g., stroke, multiple sclerosis, Parkinson's disease; clinically significant peripheral neuropathy, or complete spinal cord injury)
* Patient has uncontrolled type I or type II diabetes as defined by their routine care clinician or diabetes with peripheral nerve involvement
* Any history of any pelvic cancer
* Patient has history of other non-pelvic neoplasia within 5 years prior to enrolment, except for a cancer that was determined to be local occurrence only, such as basal cell carcinoma, or is receiving or planning to receive anti-cancer or anti-angiogenic drugs
* Patient has proven major autoimmune disease, e.g. scleroderma or immunodeficiency (including use of biologic immunomodulatory drugs at time of procedure)
* Life expectancy of less than 1 year
* Patient is a frail elderly and/or with notable clinical evidence of sarcopaenia
* Patient is not suitable for the study as determined by their routine care physician for any other reason
* Patient is enrolled in another interventional study excepting observational studies, e.g. SNM registries or in relation to disease (see below)
* Patient participation in vigorous sporting activities where these cannot be restricted for a period of 6 weeks post-implantation.

Specific urological

* Urinary tract mechanical obstruction such as urethral stricture
* Current symptomatic urinary tract infection (UTI) or more than 3 UTIs in past year
* Pure stress incontinence or mixed incontinence where the stress component overrides the urge component
* Interstitial cystitis or bladder pain syndrome as defined by either AUA or EAU guidelines
* Suspected pudendal nerve entrapment syndrome. In patients with co-existent symptoms of chronic pelvic pain and urinary incontinence, Nantes criteria will be used for screening. Patients meeting essential criteria will be excluded from the study
* Treatment of urinary symptoms with botulinum toxin therapy in the past 12 months
* Prior attempt at pudendal nerve stimulation using an implanted lead
* Treatment of urinary symptoms with tibial or sacral nerve stimulation in the past 3 months (prior experience of either before this time is permitted provided no implants remain in-situ)

Specific technical

* Patient is significantly obese (defined as BMI ≥ 35) so as to limit electrode lead placement using standard approaches
* Skin, orthopaedic or neurological anatomical limitations that could prevent successful placement of the electrode lead
* Knowledge of planned MRIs, diathermy, microwave exposure, high output ultrasonic exposure, or RF energy exposure
* Implantable neurostimulator, pacemaker or defibrillator in situ (anywhere in body including sacral and tibial)
* Subject with a documented history of allergic response to titanium, zirconia, polyurethane, epoxy, or silicone

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Adverse Device Events | 24 hours; 1 week; 4 weeks; 3 months; 6 months
  Incidence of adverse events as defined by REGULATION (EU) 2017/745(MDR) and MDCG 2020-10/1

SECONDARY OUTCOMES:
Changes in Voiding diary data | Baseline, 28 days, 3 months, 6 months
  Changes in 5 days voiding diary data including number of incontinence episodes, number of voids, number of urgency episodes
Changes in ICIQ -UI Short Form | Baseline, 28 days, 3 months, 6 months
  ICIQ-SF-UI questionnaire: is a questionnaire for evaluating frequency, severity and impact on quality of life of urinary incontinence in research and clinical practice. It is a 4 item simple questionnaire
Changes in ICIQ-OAB Quality of Life | Baseline, 28 days, 3 months, 6 months
  ICIQ-OAB Qol questionnaire: is a robust, subject-completed questionnaire for evaluating quality of life (QoL) in subjects with overactive bladder, for use in research and clinical practice. The questionnaire explores in detail the impact on subject's lives of overactive bladder and can be used as an outcome measure to assess impact of different
Changes in PGI-I | Baseline, 28 days, 3 months, 6 months
  Patient Global Impression of Improvement (PGI-I): The PGI-I is a subject-completed transition scale that is a single question asking the subject to rate their urinary tract condition now, as compared with how it was prior to before beginning treatment on a 7 point scale
Changes in FSFI | Baseline, 28 days, 3 months, 6 months
  FSFI - questionnaire: The Female Sexual Function Index (FSFI) is a widely used multidimensional self-reported questionnaire on Female Sexual Dysfunction. It consists of 19 items and assesses 6 domains, including desire, arousal, lubrication, orgasm, satisfaction and pain.
Technical Outcomes | 24 hours postoperatively
  Number of patients successfully implanted
Measurement of EMG | During procedure, 24 hours and 6 months
  Intra-operative and post-operative (ambulatory) measurements of electromyography

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Antwerp, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No